CLINICAL TRIAL: NCT02309749
Title: CAP Pilot Study for Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: FPH-AD13-01
Record Dates: First submitted 2013-04-02; First posted 2014-12-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Naive cohort
  Interventions: Other: CAP

INTERVENTIONS:
Other: CAP

SUMMARY:
This is a pilot to review the feasibility of a program that assists patients towards therapy compliance by scheduled intervention through the first month of therapy. The hypothesis of this study is that the trial program will function as intended and average patient adherence will be over 4 hours per night.

ELIGIBILITY:
Inclusion Criteria

* 21 to 75 years of age
* Diagnosed with OSA (AHI >5 events/hour) and eligible for Continuous Positive Airway Pressure (CPAP) treatment under local requirements
* Must be initiated on program (i.e. received their device) within 12 weeks of CPAP titration study
* Naïve to CPAP therapy, i.e have not been prescribed CPAP in the past
* Access to a cellphone

Exclusion Criteria:

* Contraindicated for CPAP therapy
* Medically unstable condition/diagnosis that is not yet under control
* Co-existing sleep disorder (however clinically diagnosed insomnia can be included in the study)
* Periodic Leg MOvement Arousal Index greater than 15/hr
* Home titration of longer than 5 days

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep laboratory, DME supplier
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of delivery of SMS messages to participant | 30 days
  Cross check recieved messages logged in a diary by the participant to those sent by CAP

SECONDARY OUTCOMES:
Participant CPAP Adherence | 30 nights
  Assess the adherence of participants to CPAP therapy while enrolled in CAP

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clayton Sleep Institute, St Louis, Missouri
  - Sleep Therapy Research Center, San Antonio, Texas